CLINICAL TRIAL: NCT01439373
Title: Double-Blind, Randomized, Placebo-Controlled Study to Assess Safety, Efficacy, and Pharmacokinetics (PK) of GSK2336805 in Combination With Peginterferon and Ribavirin in Treatment-naive Chronic Hepatitis C Subjects With Hepatitis C Virus Genotypes 1 or 4
Brief Title: Safety, Antiviral Activity, and Pharmacokinetics of GSK2336805 With Peginterferon and Ribavirin in Chronic Hepatitis C Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115519
Record Dates: First submitted 2011-07-07; First posted 2011-09-23 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic hepatitis C; NS5A inhibitor; ribavirin; pegylated interferon; GSK2336805
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — GSK2336805; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK2336805 (Experimental): Study Part 1
  Interventions: Drug: GSK2336805
- Placebo (Placebo Comparator): Study Part 1
  Interventions: Drug: GSK2336805 Matching Placebo
- GSK2336805 + pegylated interferon alfa-2a + ribavrin (Experimental): Study Part 2
  Interventions: Drug: GSK2336805; Drug: Pegylated interferon alfa-2a; Drug: Ribavirin
- Placebo + pegylated interferon alfa-2a + ribavirin (Active Comparator): Study Part 2
  Interventions: Drug: Pegylated interferon alfa-2a; Drug: Ribavirin; Drug: GSK2336805 Matching Placebo

INTERVENTIONS:
Drug: GSK2336805 — Active Investigational Drug
  Arms: GSK2336805; GSK2336805 + pegylated interferon alfa-2a + ribavrin
Drug: Pegylated interferon alfa-2a — Standard of Care drug
  Other Names: Pegasys
  Arms: GSK2336805 + pegylated interferon alfa-2a + ribavrin; Placebo + pegylated interferon alfa-2a + ribavirin
Drug: Ribavirin — Standard of Care drug
  Arms: GSK2336805 + pegylated interferon alfa-2a + ribavrin; Placebo + pegylated interferon alfa-2a + ribavirin
Drug: GSK2336805 Matching Placebo — Placebo of Investigational Drug
  Other Names: Placebo
  Arms: Placebo; Placebo + pegylated interferon alfa-2a + ribavirin

SUMMARY:
GSK2336805 is a hepatitis C virus (HCV) NS5A inhibitor being developed for the treatment of chronic hepatitis C (CHC). This study will assess the safety, antiviral activity, and pharmacokinetics of GSK2336805 alone and in combination with peginterferon alfa 2a and ribavirin in subjects with chronic hepatitis C (CHC).

DETAILED DESCRIPTION:
HCV infection is a major public health problem globally and a leading cause of chronic liver disease. New medications are needed that are better tolerated and offer a greater chance of achieving sustained viral clearance compared to currently available therapy. GSK2336805 is a HCV NS5A inhibitor being developed for the treatment of subjects with CHC. This Phase II, double blind, randomized, placebo-controlled study will assess the safety, antiviral activity, and pharmacokinetics of GSK2336805 alone and in combination with peginterferon alfa 2a and ribavirin in subjects with CHC. Subjects will be randomly allocated on a 2:1 basis to GSK2336805 or matching placebo and will be stratified by IL28B status and HCV viral genotype (genotype 1 or 4). The study consists of 2 parts. In Part 1, GSK2336805 or matching placebo will be given as single-dose monotherapy (Day 1). In Part 2, GSK2336805 or matching placebo will be co-administered with peginterferon alfa-2a and ribavirin through 4 weeks of treatment (Days 2 to 28). After completion of Part 2, GSK2336805/matching placebo will be discontinued and subjects will be offered continued standard-of-care anti-HCV therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented chronic genotype 1 or genotype 4 HCV infection
* Naïve to all HCV antiviral treatment(s)
* Agree to IL28B genotyping
* A body mass index >18 kg/m2 but not exceeding 36 kg/m2
* Liver biopsy obtained within 3 years (36 calendar months) prior to the Day 1 visit, with a fibrosis classification of non-cirrhotic. If no recent (<36 months) liver biopsy is available, a study qualifying biopsy must be performed prior to Baseline (Day 1)
* All fertile males and females must use two forms of effective contraception between them during treatment and during the 24 weeks after treatment ends
* Otherwise healthy as determined by the medical history, physical examination, ECG findings, and clinical laboratory measurements performed at Screening

Key Exclusion Criteria:

* Positive test at Screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody
* History of any other clinically significant chronic liver disease
* History of ascites, variceal hemorrhage, hepatic encephalopathy, or conditions consistent with decompensated liver disease
* Positive results on urine screen for drugs of abuse test at Screening (unless used as medical treatment, e.g., with a prescription)
* History of alcohol/drug abuse or dependence within 6 months of the study start (unless participating in a controlled rehabilitation program)
* Screening ECG corrected QT interval value greater than 450 ms and/or clinically significant ECG findings
* A personal or family history of Torsade de Pointes findings
* Pregnant or nursing women
* Males with a female partner who is pregnant
* Abnormal hematological and biochemical parameters as specified in the protocol
* History of major organ transplantation with an existing functional graft
* Thyroid dysfunction not adequately controlled
* Subjects with a history of suicide attempt or hospitalization for depression in the past 5 years and/or any current (within 6 months) severe or poorly controlled psychiatric disorder
* History or current evidence of immunologic disorder; pulmonary, cardiac, or pulmonary disease; seizure disorder; cancer or history of malignancy that in the opinion of the investigator makes the subject unsuitable for the study
* Participation in a clinical study with an investigational drug, biologic, or device within 3 months prior to first dose administration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07-07 (Actual); Primary Completion 2011-12-05 (Actual); Study Completion 2011-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (9):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Coronado, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Miramar, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Gardner S, Cutrell A, Elko-Simms C, Adkison K, Hamatake R, Walker J, Rodriguez-Torres M, Hong Z. A double-blind, randomized, placebo-controlled study to assess the safety, antiviral activity and pharmacokinetics of GSK2336805 when given as monotherapy and in combination with peginterferon alfa-2a and ribavirin in hepatitis C virus genotype 1-infected treatment-naive subjects. Liver Int. 2014 Jul;34(6):e89-95. doi: 10.1111/liv.12334. Epub 2013 Oct 16. PMID 24107072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 5 sites in the United States. The first participant was randomly assigned to study drug on 20 July 2011 and the last participant completed the study on 05 December 2011.
Pre-assignment Details: A total of 16 participants were enrolled and randomly assigned to study medication. One participant with genotype-1 who was randomly assigned to study medication withdrew before receiving the first dose and was not included in any of the analysis populations.
Groups:
- GSK2336805 60 mg + PEG + RIBA: Eligible participants received GSK2336805 60 milligram (mg) orally once daily on Day 1 (Part A) of the study. Part 2 of the study then proceeded without interruption with the co-administration of GSK2336805 60 mg once daily with peginterferon alfa-2a (PEG) 180 microgram (mcg) per week as subcutaneous injection (SC) and ribavirin (RIBA) 1000 mg (if <75 kilogram [kg]) or 1200 mg (if <75 kg) orally in 2 divided doses with food (morning and evening) (2 or three 200 mg tablets in the morning and three 200 mg tablets in the evening) through 4 weeks of treatment from Day 2 through Day 28 of the study.
- Placebo + PEG + RIBA: Eligible participants received matching placebo orally once daily on Day 1 (Part A) of the study. Part 2 of the study then proceeded without interruption with the co-administration of matching placebo once daily with PEG 180 mcg per week as SC and RIBA 1000 mg (if <75 kg) or 1200 mg (if <75 kg) orally in 2 divided doses with food (morning and evening) (2 or three 200 mg tablets in the morning and three 200 mg tablets in the evening) through 4 weeks of treatment from Day 2 through Day 28 of the study.
Period: Monotherapy (Day 1)
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Started | 11 | 5
Completed | 11 | 4
Not Completed | 0 | 1
Not completed — Participant Dropped-out at Day 1 visit | 0 | 1
Period: Combined With PEG and RIBA (Day 2 to 28)
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Started | 11 | 4
Completed | 9 | 4
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK2336805 60 mg + PEG + RIBA: Eligible participants received GSK2336805 60 mg orally once daily on Day 1 (Part A) of the study. Part 2 of the study then proceeded without interruption with the co-administration of GSK2336805 60 mg once daily with PEG 180 mcg per week as SC and RIBA 1000 mg (if <75 kg) or 1200 mg (if <75 kg) orally in 2 divided doses with food (morning and evening) (2 or three 200 mg tablets in the morning and three 200 mg tablets in the evening) through 4 weeks of treatment from Day 2 through Day 28 of the study.
- Total: Total of all reporting groups
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA | Total
Number analyzed (Participants) | 11 | 4 | 15
Age, Customized [Number; unit: Particiapnts]
  31 to 67 years | 11 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 10 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 3 | 2 | 5
  White - White/Caucasian/European Heritage | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Achieving Rapid Virological Response (RVR) at Day 28, Nominal Analysis
Description: RVR was defined as the proportion of participants below the assay lower limit of detection (LOD) <18 International units per milliliter (IU/mL) for Hepatitis C virus (HCV) ribonucleic acid (RNA) after 4 weeks of treatment (Day 28). Participants achieving RVR at Day 28 were considered treatment responders. Participants with missing HCV RNA values at Day 28 or discontinued before Day 28 were considered as treatment failure . Proportion of participants with HCV genotype 1 achieving RVR was the primary comparison of interest to show superiority of GSK2336805 over placebo in genotype 1 participants.
Time Frame: Day 28
Population: Intent-to-Treat Exposed population comprised of all participants who meet study criteria and were randomly assigned to treatment in the study with documented evidence of had received at least 1 dose of randomized treatment and at least 1 post-baseline HCV RNA measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  HCV RNA >= Low Limit of Quantification (LLOQ) | 3 | 3
  Undetectable HCV RNA | 8 | 1

2. Primary Outcome: Number of Participant Achieving RVR at Day 28, (Primary and Supportive Analyses)
Description: RVR was defined as the proportion of participants LOD <18 IU/mL for HCV RNA after 4 weeks of treatment (Day 28). Participants achieving RVR at Day 28 were considered treatment responders. Participants with missing HCV RNA values at Day 28 or discontinued before Day 28 were considered as treatment failure. Proportion of participants with HCV genotype 1 achieving RVR was the primary comparison of interest to show superiority of GSK2336805 over placebo in genotype 1 participants. The primary and supportive analysis differs from the nominal analysis as supportive analysis is assessed at Day 28 ± 2 (2 days visit window) whereas, the nominal analysis was assessed at Day 28.
Time Frame: Day 28
Population: Intent-to-Treat Exposed population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  Undetectable HCV RNA | 7 | 1
  HCV RNA >= LLOQ | 4 | 3

3. Primary Outcome: Probability of Participants With HCV Genotype 1 Achieving RVR At Day 28, Nominal Analysis
Description: The primary comparison of interest was performed using a Bayesian probability model. Probability of achieving undetectable HCV RNA distribution analyzed by nominal analysis was reported.
Time Frame: Day 28
Population: Intent-to-Treat Exposed population.
Measure: Mean (Standard Deviation); unit: Posterior probability
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Posterior probability | 0.67 (0.101) | 0.21 (0.064)
Statistical Analysis 1: Comparison: GSK2336805 60 mg + PEG + RIBA vs Placebo + PEG + RIBA; Test type: Other; Bayesian probability model; P1= P(p805 >pPLC +0.3 | data)= 0.905. A probability of 95% (P1 > 0.95) or greater was to be considered 'substantial evidence of superiority; Mean posterior difference = 0.46, Standard Deviation 0.119 — Posterior Distribution of Difference= p805 - pPLC, where, p805 is the RVR rate for GSK2336805 and pPLC is the RVR rate for Placebo. 95% credible set was defined as the 2.5 and 97.5 percentiles. 95% credible interval for the estimate was 0.22 to 0.68

4. Primary Outcome: Probability of Participants With HCV Genotype 1 Achieving RVR at Day 28, Primary and Supportive Analyses
Description: The primary comparison of interest was performed using a Bayesian probability model. Probability of achieving undetectable HCV RNA distribution analyzed was reported.
Time Frame: Day 28
Population: Intent-to-Treat Exposed population.
Measure: Mean (Standard Deviation); unit: Posterior probability
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Posterior probability | 0.62 (0.104) | 0.21 (0.064)
Statistical Analysis 1: Comparison: GSK2336805 60 mg + PEG + RIBA vs Placebo + PEG + RIBA; Test type: Other; Bayesian probability model; P1= P(p805 >pPLC +0.3 | data)= 0.822. A probability of 95% (P1 > 0.95) or greater was to be considered 'substantial evidence of superiority; Mean posterior difference = 0.41, Standard Deviation 0.122 — Posterior Distribution of Difference= p805 - pPLC, where, p805 is the RVR rate for GSK2336805 and pPLC is the RVR rate for Placebo. 95% credible set was defined as the 2.5 and 97.5 percentiles. 95% credible interval for the estimate was 0.17 to 0.6

5. Primary Outcome: Number of Participants With HCV Genotype 1 With Virologic Response
Description: Serum for determination of HCV genotype was collected at the screening visit. Genotype was determined by the VERSANT HCV genotype 2.0 Assay (LiPA). Number of participants with HCV genotype 1 were reported.
Time Frame: Day 7, 14 and 21
Population: Intent-to-Treat Exposed population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  Day 7, Undetectable HCV RNA | 1 | 0
  Day 7, Detectable HCV RNA but < LLOQ | 1 | 0
  Day 7, HCV RNA >= LLOQ | 9 | 4
  Day 14, Undetectable HCV RNA | 4 | 0
  Day 14, Detectable HCV RNA but < LLOQ | 2 | 0
  Day 14, HCV RNA >= LLOQ | 5 | 4
  Day 21, Undetectable HCV RNA | 7 | 0
  Day 21, Detectable HCV RNA but < LLOQ | 1 | 0
  Day 21, HCV RNA >= LLOQ | 3 | 4

6. Primary Outcome: Change From Baseline in HCV Viral Load During 24 Hour (h) Following a Single Dose of GSK2336805 on the Log 10 Scale
Description: Blood samples for determination of HCV RNA levels were collected at immediately prior to and 1, 2, 4, 6, and 8 and 24 h after the first dose in Part 1 (Day 1). Measurement of HCV viral load was analyzed by the central laboratory using the COBAS AmpliPrep/COBAS TaqMan HCV test. Baseline was defined as the last non-missing assessment on or before the first dose of study drug. Change from Baseline was computed as value at post Baseline specified time point minus Baseline value. Virus RNA levels reported as <43 are undetectable levels. If the result for HCV RNA (IU/ML) was <43, then change from Baseline was calculated using 42, and the change from Baseline on the log scale was calculated using log (42).
Time Frame: Day 1 (Baseline [Pre-dose], 1, 2, 4, 6, and 8 and 24 h)
Population: Intent-to-Treat Exposed population.
Measure: Mean (Standard Deviation); unit: Log IU/mL
Groups:
- GSK2336805 60 mg (Part A): Eligible participants received GSK2336805 60 mg once daily on Day 1 (Part A) of the study.
- Placebo (Part A): Eligible participants received matching placebo once daily on Day 1 (Part A) of the study
Arm/Group | GSK2336805 60 mg (Part A) | Placebo (Part A)
Number analyzed (Participants) | 11 | 4
Log IU/mL
  1 h post-dose | 0.02 (0.31) | -0.01 (0.06)
  2 h post-dose | -0.03 (0.21) | -0.00 (0.07)
  4 h post-dose | -0.70 (0.42) | -0.07 (0.07)
  6 h post-dose | -1.37 (0.63) | 0.08 (0.15)
  8 h post-dose | -1.83 (0.81) | 0.07 (0.11)
  24 h post-dose | -2.38 (1.15) | -0.11 (0.11)

7. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Event (SAE) During Treatment Period
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE include AEs those result in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Up to Day 28
Population: Safety population was consisted of all participants who received at least 1 dose of study medication (GSK2336805 or matching placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  Any AE | 11 | 4
  Any SAE | 0 | 0

8. Primary Outcome: Change From Baseline in QTcF Interval at Day 2 and 28
Description: Single 12-lead electrocardiogram (ECG) was obtained. The standard ECG criteria of potential clinical importance were 1) absolute QTc Interval, > 450 milliseconds (msec), 2) absolute PR Interval, <110 msec, 3) absolute QRS Interval, < 75 msec and 4) increase from baseline in QTc > 60 msec. QTc Interval was calculated using Frederica correction formula: QTcF = QT / (RR)^1/3. Change from Baseline was calculated by subtracting the Baseline assessment value from post Baseline visit value. Baseline was defined as the last non-missing assessment on or before the first dose of study drug. The change from Baseline in QTc Interval at Day 2 and 28 were reported.
Time Frame: Baseline (Day 1, Pre-dose ), Day 2 and Day 28
Population: Safety population.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
msec
  DAY 2 | 0.01 (17.921) | 0.82 (10.714)
  DAY 28: number analyzed (Participants) | 10 | 4
  DAY 28 | -5.15 (15.049) | 9.13 (9.328)

9. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post Baseline Toxicity Grade Hematology Parameters for Day 1 to Day 28
Description: Laboratory abnormalities were graded according to the modified division of AIDS ( DAIDS）version 1.0. Shift from Baseline to worst post baseline toxicity grade (where applicable) were presented for Day 1 to Day 28. The toxicity Grades were, Grade 1: mild (no or minimal interference with usual social & functional activities); Grade 2: moderate (greater than minimal interference with usual social and functional activities); Grade 3: severe (inability to perform usual social and functional activities); Grade 4: potentially life threatening (inability to perform basic self-care functions or Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death). Hematology parameters were red blood cell, hemoglobin, hematocrit, platelet white blood cell count with differential leukocyte count, mean corpuscular volume, prothrombin time and international normalized ratio.
Time Frame: Baseline (Day 1) to Day 28
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  Hemoglobin, No toxicity | 7 | 3
  Hemoglobin, Grade 1 | 3 | 1
  Hemoglobin, Grade 2 | 1 | 0
  International normalized ratio, No toxicity | 10 | 3
  International normalized ratio, Grade 1 | 1 | 1
  Lymphocytes absolute, No toxicity | 10 | 4
  Lymphocytes absolute, Grade 4 | 1 | 0
  Platelet count, No toxicity | 10 | 3
  Platelet count, Grade 1 | 1 | 0
  Platelet count, Grade 2 | 0 | 1
  Prothrombin time, No toxicity | 10 | 3
  Prothrombin time, Grade 1 | 1 | 1
  Total neutrophils, absolute, No toxicity | 7 | 2
  Total neutrophils, absolute, Grade 1 | 1 | 2
  Total neutrophils, absolute, Grade 2 | 2 | 0
  Total neutrophils, absolute, Grade 3 | 1 | 0
  White cell count, No toxicity | 8 | 3
  White cell count, Grade 1 | 2 | 1
  White cell count, Grade 2 | 1 | 0

10. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post Baseline Toxicity Grade for Serum Chemistry Parameters for Day 1 to Day 28
Description: Abnormalities were graded according to the modified DAIDS version 1.0. Shift from Baseline to worst post Baseline toxicity grade were presented for Day 1 to Day 28. The toxicity Grades were, Grade 1: mild (no or minimal interference with usual social & functional activities); Grade 2: moderate (greater than minimal interference with usual social and functional activities); Grade 3: severe (inability to perform usual social and functional activities); Grade 4: potentially life threatening (inability to perform basic self-care functions or Medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death). Clinical chemistry parameters were alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, creatine phosphokinase, total CO2, chloride, creatinine, glucose, sodium, phosphate, potassium, total albumin, total bilirubin, and direct bilirubin. Only participants with change in toxicity grades are reported.
Time Frame: Baseline (Day 1) and 28
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  Alanine aminotransferase, No toxicity | 11 | 2
  Alanine aminotransferase, Grade 1 | 0 | 1
  Albumin, No toxicity | 11 | 3
  Albumin, Grade 1 | 0 | 1
  Aspartate aminotransferase, No toxicity | 8 | 1
  Aspartate aminotransferase, Grade 1 | 1 | 1
  Aspartate aminotransferase, Grade 2 | 0 | 1
  Total Bilirubin, No toxicity | 9 | 3
  Total Bilirubin, Grade 1 | 2 | 0
  Total Bilirubin, Grade 2 | 0 | 1
  Carbon dioxide, No toxicity | 8 | 1
  Carbon dioxide, Grade 1 | 1 | 1
  Creatine phosphokinase, No toxicity | 10 | 4
  Creatine phosphokinase, Grade 1 | 1 | 0
  Glucose, No toxicity | 5 | 4
  Glucose, Grade 1 | 4 | 0
  Glucose, Grade 2 | 1 | 0
  Phosphorus, inorganic, No toxicity | 8 | 4
  Phosphorus, inorganic, Grade 1 | 2 | 0
  Phosphorus, inorganic, Grade 2 | 1 | 0
  Potassium, No toxicity | 10 | 3
  Potassium, Grade 1 | 1 | 0
  Sodium, No toxicity | 9 | 4
  Sodium, Grade 2 | 2 | 0

11. Secondary Outcome: Number of Participants With Shifts in Urinalysis Parameters From Normal at Baseline to Abnormal
Description: The urinalysis parameters analyzed were Leukocyte esterase, bilirubin, occult blood, glucose, ketones, nitrite, pH, specific gravity and dipstick assessments. Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important urinalysis findings at specified visit were reported. Visits where no abnormal values were observed not reported.
Time Frame: Day 14, 28, Follow-up (Day 42)
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants
  Occult blood, Day 14: number analyzed (Participants) | 9 | 4
  Occult blood, Day 14 | 0 | 1
  Occult blood, Follow-up: number analyzed (Participants) | 10 | 4
  Occult blood, Follow-up | 0 | 1
  Ketone, Day 14: number analyzed (Participants) | 9 | 4
  Ketone, Day 14 | 1 | 2
  Nitrate, Day 14: number analyzed (Participants) | 9 | 3
  Nitrate, Day 14 | 1 | 1
  Leukocytes, Day 14: number analyzed (Participants) | 9 | 2
  Leukocytes, Day 14 | 1 | 1

12. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern
Description: The potential clinical importance ranges (low and high) of the vital sign parameters were for systolic blood pressure (<85 and >160 millimeter of mercury [mmHg]), diastolic blood pressure (<45 and >100 mmHg) and heart rate (<40 and >110 beats per minute). Only those parameters for which at least one value of potential clinical importance was reported are summarized. The number of participants with potential clinical important vital parameter findings at any visit were reported.
Time Frame: Up to 42 days
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Participants | 0 | 0

13. Secondary Outcome: Mean Serum HCV RNA Levels at Baseline (Day 1), Day 2 and Day 28
Description: Blood samples for determination of HCV RNA levels were collected from screening, immediately prior to and 1, 2, 4, 6, and 8 h after the first dose in Part 1 (Day 1), during Part 2 on Days 2 (24 h after the Day 1 dose), 7, 14, 21, and 28, and at the post-treatment follow-up visit on Day 42. All viral load samples, with the exception of the one taken during the screening visit, were taken in duplicate. The actual time and date of each sample collection will be recorded. Measurement of HCV viral load was analyzed by the central laboratory using the COBAS AmpliPrep/COBAS TaqMan HCV test.
Time Frame: Baseline (Day 1, pre-dose), Day 2 (24 h, Post-dose) and Day 28
Population: Intent-to-Treat Exposed population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log IU/mL
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Log IU/mL
  Day 1, Pre-dose, | 6.61 (0.37) | 5.43 (0.43)
  Day 2, 24 h post-dose | 4.23 (1.41) | 5.33 (0.40)
  Day 28, Pre or Post ante meridian (AM) dose: number analyzed (Participants) | 9 | 4
  Day 28, Pre or Post ante meridian (AM) dose | 1.80 (0.45) | 3.44 (1.73)

14. Secondary Outcome: Mean Change From Baseline in Serum HCV RNA Levels at Day 2 and Day 28
Description: as for outcome 13
Time Frame: Baseline (Day 1, Pre -dose ) and Day 2 (24 h, post-dose), Day 28
Population: Intent-to-Treat Exposed population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log IU/mL
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Log IU/mL
  Day 2, 24 h post-dose | -2.38 (1.15) | -0.11 (0.11)
  Day 28, Pre or Post AM dose: number analyzed (Participants) | 9 | 4
  Day 28, Pre or Post AM dose | -4.78 (0.39) | -1.99 (1.36)

15. Secondary Outcome: Change From Baseline in Serum Alanine Aminotransferase Levels
Description: Blood samples were collected at Baseline (Day 1, Pre-dose), Day 7, 14, 21, 28 and 42 for determination of serum alanine aminotransferase levels. Baseline was defined as the last non-missing assessment on or before the first dose of study drug. Change from Baseline was computed as value at post Baseline specified time point minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 7, 14, 21, 28 and 42
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
Units per litre (U/L)
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | -15.3 (11.67) | -15.0 (21.79)
  Day 14: number analyzed (Participants) | 10 | 4
  Day 14 | -25.7 (20.80) | -0.5 (15.29)
  Day 21: number analyzed (Participants) | 10 | 4
  Day 21 | -25.9 (23.78) | -10.0 (15.34)
  Day 28: number analyzed (Participants) | 10 | 4
  Day 28 | -24.4 (22.96) | 7.0 (27.68)
  Follow-up (Day 42): number analyzed (Participants) | 10 | 4
  Follow-up (Day 42) | -19.5 (25.44) | -19.5 (12.79)

16. Secondary Outcome: Median Serum Alanine Aminotransferase at Baseline, Day 7, 14, 21, 28 and 42
Description: Blood samples were collected at Baseline (Day 1, Pre-dose), Day 7, 14, 21, 28 and 42 for determination of serum alanine aminotransferase levels.
Time Frame: Baseline (Day 1, Pre-dose), Day 7, 14, 21, 28 and 42
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: U/L
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
Number analyzed (Participants) | 11 | 4
U/L
  Baseline | 56.0 [24 to 95] | 43.5 [29 to 93]
  Day 7: number analyzed (Participants) | 10 | 3
  Day 7 | 41.5 [22 to 59] | 37.0 [29 to 53]
  Day 14: number analyzed (Participants) | 10 | 4
  Day 14 | 28.0 [20 to 44] | 48.5 [36 to 74]
  Day 21: number analyzed (Participants) | 10 | 4
  Day 21 | 27.0 [14 to 47] | 39.0 [24 to 67]
  Day 28: number analyzed (Participants) | 10 | 4
  Day 28 | 28.0 [16 to 58] | 48.0 [19 to 122]
  Follow-up (Day 42): number analyzed (Participants) | 10 | 4
  Follow-up (Day 42) | 29.0 [19 to 48] | 27.0 [20 to 57]

17. Secondary Outcome: Mean Area Under the Concentration-time Curve (AUC[0-24]), AUC From Time 0 Extrapolated to Infinity (AUC[0-inf]) of GSK2336805, at Day 1
Description: AUC values were determined using the linear-up, log-down trapezoidal rule. The individual plasma concentration and actual time data was used to derive the PK parameters of GSK2336805 on Day 1 by noncompartmental PK analyses. For the calculation of PK parameters all plasma concentrations that were below quantification limit (BLQ) before the first measurable concentration were set to zero. The BLQ values that occur at the end of the profile after the last quantifiable concentration were set to missing. Actual sampling times, rather than scheduled sampling times, were used in all computations of PK parameters.
Time Frame: 0.0 (pre-dose) and 1, 2, 4, 6, 8, and 24 h post-dose (morning of Day 2)
Population: Intensive Pharmacokinetic (PK) Population comprised of all participants who received GSK2336805, undergo intensive PK sampling during part 1 (Day 1) of the study, and provide evaluable GSK2336805 PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram (ng)*h/mL
Arm/Group | GSK2336805 60 mg (Part A)
Number analyzed (Participants) | 11
Nanogram (ng)*h/mL
  AUC (0-24) | 2977.79 (56.9)
  AUC(0-inf) | 3284.90 (61.6)

18. Secondary Outcome: Median Time of Maximal Plasma Concentration (Tmax) of GSK2336805 and Lag Time Before First Observation of Quantifiable Concentration (Tlag) at Day 1
Description: The individual plasma concentration and actual time data was used to derive the PK parameters of GSK2336805 on Day 1 by noncompartmental PK analyses. For the calculation of PK parameters all plasma concentrations that were BLQ before the first measurable concentration were set to zero. The BLQ values that occur at the end of the profile after the last quantifiable concentration were set to missing. Actual sampling times, rather than scheduled sampling times, were used in all computations of PK parameters
Time Frame: 0.0 (pre-dose) and 1, 2, 4, 6, 8, and 24 h post-dose (morning of Day 2)
Population: Intensive PK Population.
Measure: Median (Full Range); unit: h
Arm/Group | GSK2336805 60 mg (Part A)
Number analyzed (Participants) | 11
h
  Tmax | 2.00 [0.517 to 4.067]
  Tlag | 0.00 [0.00 to 0.00]

19. Secondary Outcome: Mean Maximum Plasma Concentration of GSK2336805 (Cmax) and Concentration at 24 h (C24) at Day 1
Description: The individual plasma concentration and actual time data was used to derive the PK parameters of GSK2336805 on Day 1 by non-compartmental PK analyses. For the calculation of PK parameters all plasma concentrations that were BLQ before the first measurable concentration were set to zero. The BLQ values that occur at the end of the profile after the last quantifiable concentration were set to missing. Actual sampling times, rather than scheduled sampling times, were used in all computations of PK parameters.
Time Frame: 0.0 (pre-dose) and 1, 2, 4, 6, 8, and 24 h post-dose (morning of Day 1)
Population: Intensive PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK2336805 60 mg (Part A)
Number analyzed (Participants) | 11
ng/mL
  Cmax | 404.84 (51.1)
  C24 | 26.98 (92.6)

20. Secondary Outcome: Mean Apparent Clearance (CL/F) of GSK2336805
Description: as for outcome 18
Time Frame: 0.0 (pre-dose) and 1, 2, 4, 6, 8, and 24 h post-dose (morning of Day 1)
Population: Intensive PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- GSK2336805 60 mg: Eligible participants received GSK2336805 60 mg once daily on Day 1 (Part A) of the study
Arm/Group | GSK2336805 60 mg
Number analyzed (Participants) | 11
L/h | 18.27 (61.6)

21. Secondary Outcome: Mean Pre-dose Concentration and Concentration at 2 to 4 h Post-dose of GSK2336805 at Days 7, 14, 21, and 28
Description: as for outcome 18
Time Frame: 0 (pre-dose), 0 to 2 h, > 2 h up to 4 h, > 4 h up to 6 h, or > 6 h up to 10 h on Days 7, 14, 21 and 28
Population: Sparse PK population included all participant who received GSK2336805, underwent sparse PK sampling during part 2 of the study, and provide at least one evaluable GSK2336805 PK concentration. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | GSK2336805 60 mg (Part A)
Number analyzed (Participants) | 10
ng/ml
  Day 7, Predose: number analyzed (Participants) | 2
  Day 7, Predose | 37.80 (3.16)
  Day 7, >2 to 4 h: number analyzed (Participants) | 5
  Day 7, >2 to 4 h | 621.40 (281.43)
  Day 7, >4 to 6 h: number analyzed (Participants) | 2
  Day 7, >4 to 6 h | 314.19 (2.62)
  Day 14, Predose: number analyzed (Participants) | 2
  Day 14, Predose | 121.57 (101.40)
  Day 14, >0 to 2 h: number analyzed (Participants) | 1
  Day 14, >0 to 2 h | 518.82 (NA) — Only one participant was available for analysis therefore, dispersion was not calculated.
  Day 14, >2 to 4 h: number analyzed (Participants) | 3
  Day 14, >2 to 4 h | 364.75 (86.48)
  Day 14, >4 to 6 h: number analyzed (Participants) | 3
  Day 14, >4 to 6 h | 304.03 (257.03)
  Day 21, Predose: number analyzed (Participants) | 2
  Day 21, Predose | 484.18 (610.46)
  Day 21, >2 to 4 h: number analyzed (Participants) | 3
  Day 21, >2 to 4 h | 346.00 (85.51)
  Day 21, >4 to 6 h: number analyzed (Participants) | 2
  Day 21, >4 to 6 h | 546.72 (442.29)
  Day 21, >6 to 10 h: number analyzed (Participants) | 1
  Day 21, >6 to 10 h | 317.49 (NA) — Only one participant was available for analysis therefore, dispersion was not calculated.
  Day 28, Predose: number analyzed (Participants) | 3
  Day 28, Predose | 16.95 (14.90)
  Day 28, >0 to 2 h: number analyzed (Participants) | 2
  Day 28, >0 to 2 h | 607.02 (162.62)
  Day 28, >2 to 4 h: number analyzed (Participants) | 9
  Day 28, >2 to 4 h | 402.05 (198.98)

ADVERSE EVENTS:
Time Frame: AEs were collected till end of the follow-up period (Day 42). On treatment SAE and non-SAEs were reported.
Description: Safety population was used for collection of the AEs
Arm/Group | GSK2336805 60 mg + PEG + RIBA | Placebo + PEG + RIBA
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4
Other Adverse Events (participants affected / at risk) | 11/11 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2336805 60 mg + PEG + RIBA (N=11) | Placebo + PEG + RIBA (N=4)
PYREXIA (General disorders) | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 3 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 4 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
CHILLS (General disorders) | 2 | 0
FATIGUE (General disorders) | 5 | 1
PAIN (General disorders) | 1 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
BACTERAEMIA (Infections and infestations) | 0 | 1
FOLLICULITIS (Infections and infestations) | 2 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 1
BLOOD PHOSPHORUS DECREASED (Investigations) | 1 | 0
CARBON DIOXIDE DECREASED (Investigations) | 1 | 0
HAEMATOCRIT DECREASED (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.